CLINICAL TRIAL: NCT02010125
Title: A Multi-Center Feasibility Trial Establishing Imaging and Biochemical Technologies as Measures of Knee Cartilage Composition Following Acute ACL Injury
Brief Title: Feasibility Trial Using Imaging and Biochemical Technologies to Measure Knee Cartilage Composition in Acute ACL Injury
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AFstudy
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Acute Injury of Anterior Cruciate Ligament
Keywords: Anterior Cruciate Ligament (ACL); Magnetic Resonance Imaging (MRI); Osteoarthritis (OA); Bio-specimens; Acute ACL Injury; Arthritis Foundation (AF)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, Whole Blood, Synovial Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ACL injury: Subjects with acute ACL injury will be recruited and enrolled within 28 days of injury Serum, urine, and synovial fluid will be collected at baseline, 6wks post-injury or post-surgery, 6 months, and 1 year Patients will have a quantitative MRI on both knees 7 days after initial visit, then at 6 months and 1 year.
  Patients may or may not opt for ACL reconstruction Patients will have functional testing (One-legged hop tests and Star excursion balance test) at 6 months and 1 year Patients will fill out questionnaires (Knee Osteoarthritis Outcome Survey, Veteran Rand-12, Lysholm, International Knee Documentation Committee, Marx Questionnaire) at baseline, 6 weeks, 6 months, and 1 year

SUMMARY:
This study will evaluate the bio-mechanical and biochemical abnormalities in acute ACL-injured knees over time. Data will be collected through advanced quantitative MR imaging, functional testing, and bio-specimen collection. Researchers will collect this data from the time of baseline visit, which is within 28 days of injury, through the temporal sequence of post-operative or post-injury recovery and return to activity.

The hypotheses for this study are (1) that T1ρ and T2 will be significantly elevated in the lateral side of ACL-injured knees immediately after injury (indicating damage caused by initial injury), and will not fully recover at 6-month, 1-year follow ups; (2) that T1ρ and T2 will be significantly elevated in the medial side of ACL-injured knees at 1-year follow-up; and (3) that differences in the bio-marker expression patterns can be correlated with the initial MRI findings, which would provide information regarding the full spectrum of intra-articular pathology and the subsequent clinical outcomes.

DETAILED DESCRIPTION:
This prospective longitudinal study will evaluate the biomechanical and biochemical abnormalities in acute ACL-injured and reconstructed knees through advanced quantitative MR imaging, bio-specimen collection, and functional testing.

Researchers will recruit and retain patients with acute ACL tears within 28 days of injury, and follow them longitudinally at 6 weeks, 6 months, and 12 months. Standard of Care MR imaging will be captured at baseline, then a quantitative morphological MRI and quantitative T1ρ and T2 imaging of the injured and contra-lateral knees will be taken within 7 days of baseline, and again at 6 months, and 1 year post-injury or post-surgery. Scans will not take place immediately after surgery because we are not attempting to study the immediate effect of ACL reconstruction. The physical performance testing will not be acquired until 6 months follow-up because patients will have unstable knees.

For the 6 healthy volunteers, only an MRI of the right knee will be required at 4 time points - baseline, 6 months, 12 months, and 18 months. The control volunteers will be used as a measure of reproducibility. The control volunteers will not perform any physical performance testing or study questionnaires. The purpose of the six control subjects is to track the reproducibility and physiologic variation in T1p and T2 values in a normal knee. These subjects will complete imaging at four time points, spaced six months apart. The results will help evaluate the expected range of differences in knees without a traumatic injury. This information will assist in the interpretation of values from the patients with ACL injuries as to if any observed variation is outside the expected magnitude for a healthy individual. The control subjects will also help monitor for any changes in the scanner reliability at our site and compared to the other two clinical sites. Phantoms will be scanned each month to aid in this process, and control subjects will add and help ensure that data collection is constant over time.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature subjects with age 13 - 70 years
* Sustain an acute full ACL rupture in one knee < 28 day
* May or may not undergo ACL reconstruction
* Low grade injury to the collateral ligaments not resulting in instability and not requiring reconstruction will be included

Exclusion Criteria:

* Radiographic evidence of early osteoarthritis, defined as Grade 1 joint space narrowing or Grade 1 osteophyte formation
* Injuries to other ligaments requiring surgical intervention
* Have cartilage resurfacing procedures performed at the time of injury
* Inability to undergo the standard pre- and post-injury/operative rehabilitation
* Varus or valgus instability requiring ligament repair or reconstruction (from clinical exam at time of injury)
* History of osteoarthritis and inflammatory arthritis
* Women who are pregnant are excluded
* Previous injury and/or surgery on either knee

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men and Women with acute ACL injury (within 28 days)
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Follow patients with acute ACL tears longitudinally using advanced, quantitative morphological MR imaging. | Baseline - 12 months
  Patients who are within 28 days of injury will be recruited in order to capture the acute phase of injury. Quantitative morphological MRI and quantitative T1p and T2 imaging of the injured and contra-lateral knees will be captured at their baseline visit (within 7 days of initial visit), and then again at 6 months and 12 months. The aim is to investigate longitudinal changes in cartilage matrix in ACL-injured and reconstructed knees using T1ρ and T2. We hypothesize that T1ρ and T2 will be significantly higher in defined sub-compartments of injured knees compared to the contralateral un-injured knees at baseline and follow-ups. Meniscus, ligamentous and cartilage abnormalities will be graded using MRI for correlation with cartilage T1ρ and T2.

SECONDARY OUTCOMES:
Collect and store bio-specimens | Baseline - 12 months
  Blood, urine, and synovial fluid will be collected from patients at each time point (initial visit; surgery (if applicable); 6 weeks post-injury (or post-surgery, if applicable), 6 months, and 12 months). The aim is to collect, freeze, and store these samples from each time point to develop a repository of bio-specimens, which can be correlated with imaging, clinical and functional outcomes at a later phase when funding becomes available for such assays. The hypothesis is that differences in the bio-marker expression patterns can be correlated with the initial MRI findings, which provide information regarding the full spectrum of intra-articular pathology, and the subsequent clinical outcomes.
Functional Assessments | 6 months, 12 months
  Physical performance and functional testing will only be preformed at 6 months and 1-year, and not during the initial visits due to functional limitations. Subjects will perform the "One-Legged Hop Tests" and the "Star Excursion Balance Test (SEBT)". The aim of the functional testing is to demonstrate the feasibility of relating the MRI derived morphological and biochemical measures to clinical and functional assessments.
Patient-Reported Questionnaires | Baseline - 12 months
  In addition to demographic data, the activity level of all subjects will be evaluated using the Lysholm questionnaire. Pre- and post-injury/post-operative SF-36 and IKDC evaluations will be performed to document the patient's objective and subjective complaints. Knee Injury and Osteoarthritis Outcome Score (KOOS), which is specifically used for knee injuries that result in post-traumatic OA, will be evaluated in all subjects, including 5 subscales: pain, other symptoms, function in daily living ADL, function in sports and recreation, and knee-related quality of life. The aim is to demonstrate the feasibility of relating the longitudinally acquired, novel imaging measures to the clinical outcomes as assessed by patient-reported questionnaires, and assess the magnitude and types of OA features developed over time at multiple centers.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbong B Ma, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Orthopaedic Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided at this point. If there are any queries, can contact at maben@ucsf.edu